CLINICAL TRIAL: NCT06239324
Title: Evaluation of Latanoprost Combined With Fractional Erbium- YAG Laser Versus Microneedling in Alopecia Areata Treatment
Brief Title: Evaluation of Latanoprost Combined With Fractional Erbium- YAG Laser
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Maha Nabil
Record Dates: First submitted 2024-01-16; First posted 2024-02-02 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fractional Erbium laser Technique (Group A) (Active Comparator): About 35 patients with alopecia areata will Subject to fractional Erbium (Er-YAG) laser (Fotona Xs dynamics,Slovenia) with energy of 600 mj in short pulse mode (MSP) with spot size of 7 mm diameter, frequency of 3 Hz and pixel 3. Latanoprost( xalatan 0.005% ) is applied to the treated area for all participants.
  Interventions: Drug: Latanoprost
- Micro needling Technique (Group B) (Active Comparator): About 35 patients with alopecia areata will Subject to micro needling using electronic dermapen device (Dr Pen Derma PenUltima A6) which has a disposable head personalized for each patient and sterilized after each session. the dermapen will penetrate the skin with depth 0.6 mm. It will pass vertically over the affected area in a circular pattern until pinpoint bleeding appears. Latanoprost ( xalatan 0.005% ) is applied to the treated area for all participants.
  Interventions: Drug: Latanoprost

INTERVENTIONS:
Drug: Latanoprost — Comparing between Erbium YAG laser assisted drug delivery of latanoprost versus transepidermal latanoprost delivery by microneedling in alopecia areata treatment for all participants.
  Other Names: fractional Erbium- YAG laser

SUMMARY:
Alopecia areata (AA) an autoimmune disorder of hair follicles results in varying degrees of scalp, facial and body hair loss.

Clinically, patients' presentation varies from patchy circumscribed scalp involvement to total body and scalp hair loss affects up to 2% of the general population.

The exact pathobiology of AA has still remained elusive, while the common theory is the collapse of the immune privilege of the hair follicle caused by immunological mechanism. Multiple genetic, environment factors and psychological stress contribute to the pathogenesis of Alopecia Areata .

Recent insights into the pathogenesis of AA have led to the development of new treatment strategies, such as Janus kinase inhibitors, biologics and several small molecular agents. In addition, modern therapies for AA, including antihistamines, platelet-rich plasma injection

DETAILED DESCRIPTION:
Latanoprost is a prostaglandin analogue with well-established efficacy in the treatment of open-angle glaucoma and ocular hypertension.

Make an increase in the number, thickness and length of eyelashes is an important side effect of latanoprost eye drop. This study aimed to evaluate the effect of hypertrichosis property of latanoprost in the treatment of scalp Alopecia Areata.

Numerous techniques and agents such as microneedling, dermabrasion, radiofrequency and lasers have been used to increase penetration within an approach known as transdermal drug delivery.

One of these techniques is laser-assisted drug delivery (LADD), which often uses ablative fractional lasers (CO2 or erbium: YAG lasers) because of their capacity to produce microscopic ablated channels.

LADD is a promising technique that enhances the absorption of topical molecules while adding the synergic effect.

Microneedling is a form of therapy that utilizes instruments that contain rows of thin needles that penetrate the dermis to uniform depth, creating a controlled skin injury.

Transcutaneous drug delivery via fractional laser and microneedling is a promising modality with preliminary evidence for increased hair regrowth over topical therapy alone.

Trichoscopy is a noninvasive procedure performed in dermatology clinics and is a helpful tool in determining the correct diagnosis of hair loss presentations. The five most characteristic trichoscopic findings in AA are yellow dots, black dots, broken hairs, short vellus hairs and tapering hairs. Also trichoscopy is a useful tool that allows monitoring of response during treatment of AA.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes with localized stable alopecia areata of the scalp of 3 months duration at least.

Exclusion Criteria:

1. Acute or chronic infections.
2. Pregnant or lactating women.
3. Scarring alopecia.
4. Alopecia totalis , Alopecia universalis and ophiasis.
5. Autoimmune dermatological diseases.

Ages: 30 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-04-20 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
fractional Erbium YAG laser | from baseline to 3 months after the fractional Erbium YAG laser treatment day.
  The Number of Participants With Treatment of fractional Erbium YAG laser assisted delivery of latanoprost versus micro needling with trans-epidermal latanoprost delivery to induce hair growth in alopecia areata.

CONTACTS AND LOCATIONS:
Overall Officials: Soheir AbdelHamid Ali, Assist. Prof., Principal Investigator — Department of dermatology , Venerolgy and Andrology Faculty of Medicine Qena university
Locations (1):
- Qena Hospital, Qina, Egypt

IPD SHARING:
Plan to Share IPD: No